CLINICAL TRIAL: NCT03187054
Title: Preoperative POPQ Versus Simulated Apical Support as a Guideline for Anterior or Posterior Repair at the Time of Transvaginal Apical Suspension
Brief Title: POPQ Versus Simulated Apical Support as a Guideline for Anterior or Posterior Repair During Vaginal Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Myung Jae Jeon, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUH-1705-062-853
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POPQ-based surgery (Active Comparator): will undergo anterior or posterior colporrhaphy for all of anterior or posterior vaginal prolapse stage 2 or greater (i.e. point Ba or Bp ≥-1 on the POPQ examination)
  Interventions: Procedure: anterior or posterior colporrhaphy
- Simulated apical support-based surgery (Experimental): will undergo anterior or posterior colporrhaphy only for the prolapse unresolved under simulated apical support (i.e. point Ba or Bp ≥-1 under simulated apical support)
  Interventions: Procedure: anterior or posterior colporrhaphy

INTERVENTIONS:
Procedure: anterior or posterior colporrhaphy — will be performed in a traditional manner with midline plication of the fibromuscular layer using 2-0 delayed absorbable sutures.

SUMMARY:
The objective of the Preoperative Pelvic Organ Prolapse Quantification (POPQ) versus Simulated Apical Support as a Guideline for Anterior or Posterior Repair at the Time of Transvaginal Apical Suspension (PREPARE) trial is to compare surgical outcomes of POPQ-based surgery with simulated apical support-based surgery for anterior or posterior vaginal wall prolapse at the time of transvaginal apical suspension.

DETAILED DESCRIPTION:
The PREPARE trial is a prospective, randomized trial conducted with the aim to determine non-inferiority of the primary outcome between POPQ-based surgery and simulated apical support-based surgery for anterior or posterior vaginal wall prolapse. Participants will undergo transvaginal surgery for prolapse, including the assigned procedure for anterior or posterior vaginal prolapse under general or spinal anesthesia. Concomitant procedures will be performed as intended prior to surgery. Women with a uterus in situ will undergo hysterectomy and all women will receive transvaginal vault suspension, including uterosacral ligament suspension, sacrospinous ligament fixation, and iliococcygeal suspension with both delayed absorbable and permanent sutures, according to the preference of surgeon. Incontinence surgery will also be performed for women with documented urodynamic stress incontinence.

A standardized protocol for enrollment, treatment and data collection will be employed by all sites. The study will be a single-blind study, as it is impossible to blind the study surgeon for the surgical procedure to which the subject in assigned. However, it is our intent that when feasible and ethical, all outcomes assessors and the subjects will be blinded to the treatment assignment. Postoperative follow-up will take place after 5 weeks and 6, 12, and 24 months. Patients will undergo a standard gynecological examination including POPQ and fill in questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* POPQ stage 2-4 prolapse
* Descent of vaginal apex or cervix at least ½ way into vaginal canal (i.e. POPQ point C ≥ -TVL/2)
* Correction of either anterior or posterior vaginal wall prolapse under simulated apical support (i.e. from stage 2 or greater to stage 0 or 1)
* Vaginal bulge symptoms (i.e. an affirmative response to the question 3 from the PFDI-20)
* Vaginal reconstructive surgery is planned, including a vaginal apical suspension procedure

Exclusion Criteria:

* Large pelvic mass
* Previous prolapse surgery
* Known malignancy
* Two or more inpatient hospitalizations for medical comorbidities in the previous year
* Subject wishes to retain her uterus
* Subject is unable and unwilling to participate in

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical success at 2 years after surgery | From date of surgery until the date of first documented failure, assessed up to 2 years after surgery
  surgical success is defined as the absence of all of the following criteria: (1) anterior or posterior vaginal descent beyond the hymen (i.e., point Ba or Bp >0); (2) descent of the vaginal apex beyond the half-way point of vagina (i.e., point C > -1/2×total vaginal length); (3) vaginal bulge symptoms; (4) re-treatment for prolapse by either surgery or pessary.

SECONDARY OUTCOMES:
Rate of anterior or posterior colporrhaphy | At date of surgery
  rate of anterior or posterior colporrhaphy performed during surgery
Change of POPQ values | From baseline to 2 years after surgery
  point Ba, C, Bp and TVL
Change of PFDI-20 scores | From baseline to 2 years after surgery
  the PFDI-20 is a valid and reliable condition-specific quality-of-life questionnaires for women with pelvic floor disorders. It has 20 items and 3 scales (Pelvic Organ Prolapse Distress Inventory, Colorectal-Anal Distress Inventory and Urinary Distress Inventory). Each scale is scored from 0 to 100; higher scores indicate greater symptom burden. The PFDI-20 total score is obtained by adding the scores from the 3 scale scores together (0-300).
Change of pelvic floor impact questionnaire (PFIQ-7) scores | From baseline to 2 years after surgery
  the PFIQ-7 is a valid and reliable condition-specific quality-of-life questionnaires for women with pelvic floor disorders. It has 7 questions and each question has 3 separate responses (one for each of 3 scales; Urinary Impact Questionnaire, Colo-rectal-anal Impact Questionnaire, and Pelvic Organ Prolapse Impact Questionnaire). Each scale is scored from 0 to 100; higher scores indicate greater symptom burden. The PFIQ-7 total score is obtained by adding the scores from the 3 scales together (0-300).
Change of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ)-12 scores | From baseline to 2 years after surgery
  the PISQ-12 is a valid and reliable condition-specific questionnaire that evaluates sexual function in women with urinary incontinence and/or pelvic organ prolapse. It has 12 items and responses are graded on a five-point Likert scale ranging from 0 to 4. A total of 48 is the maximum score; higher scores indicate better sexual function.
Operating times | At date of surgery
  mean or median minutes of operating times
Estimated blood loss | At date of surgery
  mean or median mililiters of estimated blood loss
Length of hospital stay | From date of admission to date of discharge, estimated average 4 days
  mean or median days of hospital stay
Rate of adverse events | From date of surgery to 2 years after surgery
  rate of cardiovascular, pulmonary, gastrointestinal, genitourinary, and neurological complications

CONTACTS AND LOCATIONS:
Overall Officials: Myung Jae Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Myung Jae, Jeon, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jeon MJ, Kim CH, Cho HH, Suh DH, Kim SR. Preoperative POPQ versus Simulated Apical Support as a Guideline for Anterior or Posterior Repair at the Time of Transvaginal Apical Suspension (PREPARE trial): study protocol for a randomised controlled trial. BMJ Open. 2020 Jan 6;10(1):e034170. doi: 10.1136/bmjopen-2019-034170. PMID 31911524